CLINICAL TRIAL: NCT00370162
Title: Safety Dermatological Evaluation: Acceptability With Gynecological Follow up - Dermacyd Delicata New Fragrance
Brief Title: Acceptability Dermacyd Delicata - New Fragrance - Lactoserum - Hygiene
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACTO_L_01839
Record Dates: First submitted 2006-08-29; First posted 2006-08-30 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Hygiene
MeSH Terms: interventions — lactoserum

INTERVENTIONS:
Drug: lactoserum

SUMMARY:
The purpose of this study is to demonstrate the safety of the gynaecological formulation in normal and usual usage condition.

ELIGIBILITY:
Inclusion Criteria:

* Integral skin in the tested region

Exclusion Criteria:

* Pregnancy or breastfeeding women
* Use of antiinflammatory or immunosuppression drugs
* Topical medication use at the tested region
* Active cutaneous gynaecological disease
* Personal history of allergic disease at the area to be treated
* Allergic or atopic history

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2006-06

PRIMARY OUTCOMES:
Adverse Events and its association with the drug in study

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, São Paulo, Brazil